CLINICAL TRIAL: NCT07335549
Title: Effect of Laparoscopic Sleeve Gastrectomy on Blood Isthmın Levels: A Prospective Cohort Study
Brief Title: Istmin Levels in Laparoscopik Sleeve Gastrectomy
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Mehmet Buğra Bozan, Proefessor, Associate MD, Saglik Bilimleri Universitesi
Other Study IDs: EFSCH1
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Obesity & Overweight; Sleeve Gastrectomy; Adipokines
Keywords: Severe Obesity; Laparoscopic Sleeve Gastrectomy; Isthmin; Adipokines
MeSH Terms: conditions — Obesity; Overweight; Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Preoperative rotuine blood samples and postopoperastive third month routine control's blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Laparoscopic Sleeve Gastrectomy Patients for Severe Obesity: Laparoscopic Sleeve Gastrectomy Patients for Severe Obesity
  Interventions: Diagnostic Test: Preoperative Serum Isthmin Levels; Diagnostic Test: Postoperative Third Month's Serum Isthmin Levels; Other: Preoperative BMI; Other: Postoperative BMI

INTERVENTIONS:
Diagnostic Test: Preoperative Serum Isthmin Levels — Preoperative Serum Isthmin Levels
Diagnostic Test: Postoperative Third Month's Serum Isthmin Levels — Postoperative Third Month's Serum Isthmin Levels
Other: Preoperative BMI — Preoperative the height and the weight of the patient will record. After that BMI will be calculated as formula "The Body Weight (kg)/(The Height (meters)x The Height (meters))
Other: Postoperative BMI — Postoperative third month's the height and the weight of the patient will record. After that BMI will be calculated as formula "The Body Weight (kg)/(The Height (meters)x The Height (meters))

SUMMARY:
Obesity is a multifactorial disease which has become a public health problem with increasing frequency, especially in recent years. Obesity causes many health problems with its negative effects on organs, systems, and psychosocial status. It is a serious risk factor for many diseases and also causes a significant increase in morbidity and mortality in these diseases.

Although dietary treatments and medical treatment options are frequently used, surgical options are still the most effective treatment. Bariatric and metabolic surgical techniques are frequently applied, especially in patients with advanced obesity and obesity-related comorbidities. The most commonly applied bariatric metabolic surgical techniques, as in our clinic, are laparoscopic sleeve gastrectomy (LSG) and Roux-en-y gastric bypass procedures.

The role of adipokines, secreted from adipose tissue and thought to play a role in the development of obesity, is quite important in the obesity mechanism, as they are effective not only in energy processes but also in metabolic processes. These adipokines secreted by adipose tissue play an active role in many mechanisms in the body, including vasoactivity, oxidative processes, immunity, lipid and glucose metabolism. Adipokines function actively in many target organs such as the pancreas, liver, and brain.

Isthmin, a relatively new adipokine expressed from brown and white adipocytes, also affects many systems like other adipokines. Studies have shown that Isthmin plays an active role in glucose and lipid metabolism, and it has been reported to play a role in many metabolic processes, from insulin resistance to hepatic steatosis.

The aim of this study is to investigate whether isthmin levels change before and after surgery in patients undergoing LSG for severe obesity, given that isthmin is thought to be associated with obesity and insulin resistance, particularly by affecting the appetite center in metabolism.

DETAILED DESCRIPTION:
Obesity is a multifactorial disease caused by genetic, environmental, and psychiatric factors. Having existed for hundreds of years, obesity has become a public health problem with increasing frequency, especially in recent years. According to WHO data, in 2016 there were 1.9 billion overweight and 650 million obese patients worldwide, and in 2022, there were 2.5 billion overweight and 890 million obese patients. This massive increase in obesity incidence in such a short time highlights that obesity is a very serious problem worldwide. According to this data, approximately 43% of the adult population over 18 years of age is overweight. This data reiterates the fact that obesity is a widespread problem with a rapidly increasing trend globally.

Obesity causes many health problems with its negative effects on organs, systems, and psychosocial status. It is a serious risk factor for many diseases and also causes a significant increase in morbidity and mortality in these diseases. Studies estimate that approximately 5 million people die worldwide due to non-communicable diseases such as cardiovascular diseases, diabetes, cancer, neurological disorders, chronic respiratory diseases, and digestive disorders related to obesity.

Today, many treatment methods are available for obesity. Although dietary treatments and medical treatment options are frequently used, surgical options are still the most effective treatment. Bariatric and metabolic surgical techniques are frequently applied, especially in patients with advanced obesity and obesity-related comorbidities. For this purpose, numerous bariatric metabolic surgical techniques have been developed. Currently, the most commonly applied bariatric metabolic surgical techniques, as in our clinic, are laparoscopic sleeve gastrectomy (LSG) and Roux-en-y gastric bypass procedures.

The role of adipokines, secreted from adipose tissue and thought to play a role in the development of obesity, is quite important in the obesity mechanism, as they are effective not only in energy processes but also in metabolic processes. These adipokines secreted by adipose tissue play an active role in many mechanisms in the body, including vasoactivity, oxidative processes, immunity, lipid and glucose metabolism. They exert their effects through paracrine and autocrine pathways. Adipokines function actively in many target organs such as the pancreas, liver, and brain.

Isthmin, a relatively new adipokine expressed from brown and white adipocytes, also affects many systems like other adipokines. Studies have shown that Isthmin plays an active role in glucose and lipid metabolism, and it has been reported to play a role in many metabolic processes, from insulin resistance to hepatic steatosis.

The aim of this study is to investigate whether isthmin levels change before and after surgery in patients undergoing LSG for severe obesity, given that isthmin is thought to be associated with obesity and insulin resistance, particularly by affecting the appetite center in metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Being diagnosed with severe obesity
* Patients who do not wish to participate in the study

Exclusion Criteria:

* Patients under 18 years of age
* Overweight patients with a Body Mass Index <40 kg/m2 and no comorbidities
* Patients with rheumatological diseases (rheumatoid arthritis, SLE, etc.)
* Patients with chronic kidney and liver failure
* Patients diagnosed with Diabetes Mellitus
* Patients with malignancy
* Patients who do not wish to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: BMI > 40 kg/m2 without comorbidity who are planned for Laparoscopic Sleeve Gastrectomy
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Serum Isthmin Levels' change | Preoperative and postoperative third month
  Serum Isthmin Levels' change

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet B Bozan, Professor, Study Director — Turkish Health Sciences University Elazig City Hospital
Locations (1):
- Elazig Fethi Sekin City Hospital, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopez-Yus M, Casamayor C, Soriano-Godes JJ, Borlan S, Gonzalez-Irazabal Y, Garcia-Sobreviela MP, Garcia-Rodriguez B, Del Moral-Bergos R, Calmarza P, Artigas JM, Lorente-Cebrian S, Bernal-Monterde V, Sanz-Paris A, Arbones-Mainar JM. Isthmin-1 (ISM1), a novel adipokine that reflects abdominal adipose tissue distribution in individuals with obesity. Cardiovasc Diabetol. 2023 Dec 8;22(1):335. doi: 10.1186/s12933-023-02075-0. PMID 38066623
- [Background] Dunmore SJ. Of fat mice and men: the rise of the adipokines. J Endocrinol. 2013 Jan 2;216(1):E1-2. doi: 10.1530/JOE-12-0513. Print 2013 Jan. No abstract available. PMID 23160965
- [Background] Fasshauer M, Bluher M. Adipokines in health and disease. Trends Pharmacol Sci. 2015 Jul;36(7):461-70. doi: 10.1016/j.tips.2015.04.014. Epub 2015 May 25. PMID 26022934
- [Background] Peri K, Eisenberg M. Review on obesity management: bariatric surgery. BMJ Public Health. 2024 Nov 27;2(2):e000245. doi: 10.1136/bmjph-2023-000245. eCollection 2024 Dec. PMID 41201062
- [Background] Kirkil C, Aygen E, Korkmaz MF, Bozan MB. QUALITY OF LIFE AFTER LAPAROSCOPIC SLEEVE GASTRECTOMY USING BAROS SYSTEM. Arq Bras Cir Dig. 2018 Aug 16;31(3):e1385. doi: 10.1590/0102-672020180001e1385. PMID 30133677
- [Background] GBD 2019 Risk Factors Collaborators. Global burden of 87 risk factors in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1223-1249. doi: 10.1016/S0140-6736(20)30752-2. PMID 33069327
- [Background] Jiang Z, Zhao M, Voilquin L, Jung Y, Aikio MA, Sahai T, Dou FY, Roche AM, Carcamo-Orive I, Knowles JW, Wabitsch M, Appel EA, Maikawa CL, Camporez JP, Shulman GI, Tsai L, Rosen ED, Gardner CD, Spiegelman BM, Svensson KJ. Isthmin-1 is an adipokine that promotes glucose uptake and improves glucose tolerance and hepatic steatosis. Cell Metab. 2021 Sep 7;33(9):1836-1852.e11. doi: 10.1016/j.cmet.2021.07.010. Epub 2021 Aug 3. PMID 34348115